CLINICAL TRIAL: NCT03447652
Title: A Randomized Controlled Trial Investigating The Effects Of A 4-Week Ankle Rehabilitation Program On High School Athletes With Chronic Ankle Instability
Brief Title: A Study Investigating The Effects Of An Ankle Rehabilitation Program On High School Athletes With Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: National Athletic Trainers' Association Research & Education Foundation (NATA Foundation) (Other)
Responsible Party: Principal Investigator, Mary Spencer Cain, Doctoral Candidate, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CON006264
Record Dates: First submitted 2018-01-28; First posted 2018-02-27 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Chronic Ankle Instability; Ankle Sprains; Ankle Rehabilitation
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: 4 independent groups
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor is blinded to which group the subjects were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): Each patient in the control group did not perform any rehabilitation exercises. Over the intervention time frame, the patient was required to check in with a member of the research team each week to discuss any changes in their ankle or report any injury incidence.
- Resistance Band Group (Experimental): Each session, patients completed resistance training using a resistance band in 4 directions of ankle motion (plantarflexion, dorsiflexion, inversion and eversion). Patients would complete 3 sets of 10 repetitions during each session. Every 3 sessions, the band resistance would increase.
  Interventions: Other: Resistance Band Ankle Rehabilitation
- Biomechanical Ankle Platform System (Experimental): The Biomechanical Ankle Platform System board is an oval shaped board that utilizes a half-sphere on the bottom of the board to allow the patient to train on an unstable surface. A one legged stance on their involved limb was performed on the Biomechanical Ankle Platform System board while clockwise and counterclockwise circles were completed. The initial rotation of direction was selected by the patient and changed every 10 seconds of the 40-second trial. Five 40-second trials were completed with 1-minute rest intervals in between the trials. Progression was determined by the supervising clinician and was based on the patient's ability to make smooth transitions between direction changes and completion of smooth circular rotations in both directions.
  Interventions: Other: Biomechanical Ankle Platform System Rehabilitation
- Combination Group (Experimental): Patients completing the combination protocol completed both the resistance band and Biomechanical Ankle Platform System board protocols during each session. The order of exercise completion was counterbalanced for each session.
  Interventions: Other: Combination Rehabilitation

INTERVENTIONS:
Other: Resistance Band Ankle Rehabilitation — Resistance Band - uses a tension band to provide resistance during ankle motion
  Arms: Resistance Band Group
Other: Biomechanical Ankle Platform System Rehabilitation — Biomechanical Ankle Platform System Board Group - uses different levels of half spheres to increase the amount of motion allowed at the ankle.
  Arms: Biomechanical Ankle Platform System
Other: Combination Rehabilitation — Combination Group - includes both the resistance band and Biomechanical Ankle Platform System programs.
  Arms: Combination Group

SUMMARY:
A randomized controlled trial investigating the effects of a 4-week ankle rehabilitation program on high school athletes with chronic ankle instability.

DETAILED DESCRIPTION:
A randomized controlled trial investigating the effects of a three different 4-week ankle rehabilitation programs on high school athletes with chronic ankle instability. We will use questionnaires to assess subjective level of function and clinical measures to assess clinical functionality via static and functional balance.

ELIGIBILITY:
Inclusion Criteria:

* active for at least 1.5 hours a week, a history of at least 1 significant ankle sprain that required medical intervention, repeated symptoms of pain, swelling, weakness, instability, and repeated episodes of "giving way".

Exclusion Criteria:

* presence of any current lower extremity injury (diagnosed by a medical professional within last 3 months with present symptoms), previous surgery to either leg, diagnosed ankle sprain within the past 6 weeks, history of ankle fractures and/or dislocations.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Static Balance Assessments | 4 weeks
  Static Balance Clinical Tests
Functional Balance Assessments | 4 weeks
  Functional Balance Clinical Tests
Patient Self-reported Outcomes | 4 to 12 weeks
  Subjective Patient Reported Outcome Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Goerger, PhD, Study Director — Georgia State University
Locations (7):
- United States (7):
  - Holy Innocents' Episcopal School, Atlanta, Georgia
  - The Lovett School, Atlanta, Georgia
  - The Westminister Schools, Atlanta, Georgia
  - Woodward Academy, College Park, Georgia
  - Decatur High School, Decatur, Georgia
  - The Walker School, Marietta, Georgia
  - Walton High School, Marietta, Georgia

IPD SHARING:
Plan to Share IPD: No
No individual participant data is planned to be shared with other researchers.

REFERENCES:
- [Background] Leininger RE, Knox CL, Comstock RD. Epidemiology of 1.6 million pediatric soccer-related injuries presenting to US emergency departments from 1990 to 2003. Am J Sports Med. 2007 Feb;35(2):288-93. doi: 10.1177/0363546506294060. Epub 2006 Nov 7. PMID 17092927
- [Background] Waterman BR, Owens BD, Davey S, Zacchilli MA, Belmont PJ Jr. The epidemiology of ankle sprains in the United States. J Bone Joint Surg Am. 2010 Oct 6;92(13):2279-84. doi: 10.2106/JBJS.I.01537. PMID 20926721
- [Background] Anandacoomarasamy A, Barnsley L. Long term outcomes of inversion ankle injuries. Br J Sports Med. 2005 Mar;39(3):e14; discussion e14. doi: 10.1136/bjsm.2004.011676. PMID 15728682
- [Background] Hertel J. Functional Anatomy, Pathomechanics, and Pathophysiology of Lateral Ankle Instability. J Athl Train. 2002 Dec;37(4):364-375. PMID 12937557
- [Background] Hiller CE, Kilbreath SL, Refshauge KM. Chronic ankle instability: evolution of the model. J Athl Train. 2011 Mar-Apr;46(2):133-41. doi: 10.4085/1062-6050-46.2.133. PMID 21391798
- [Background] Gribble PA, Delahunt E, Bleakley C, Caulfield B, Docherty CL, Fourchet F, Fong D, Hertel J, Hiller C, Kaminski TW, McKeon PO, Refshauge KM, van der Wees P, Vicenzino B, Wikstrom EA. Selection criteria for patients with chronic ankle instability in controlled research: a position statement of the International Ankle Consortium. J Orthop Sports Phys Ther. 2013 Aug;43(8):585-91. doi: 10.2519/jospt.2013.0303. Epub 2013 Jul 31. PMID 23902805
- [Background] Wikstrom EA, Hubbard-Turner T, McKeon PO. Understanding and treating lateral ankle sprains and their consequences: a constraints-based approach. Sports Med. 2013 Jun;43(6):385-93. doi: 10.1007/s40279-013-0043-z. PMID 23580392
- [Background] Harrington KD. Degenerative arthritis of the ankle secondary to long-standing lateral ligament instability. J Bone Joint Surg Am. 1979 Apr;61(3):354-61. PMID 429402
- [Background] Hintermann B, Boss A, Schafer D. Arthroscopic findings in patients with chronic ankle instability. Am J Sports Med. 2002 May-Jun;30(3):402-9. doi: 10.1177/03635465020300031601. PMID 12016082
- [Background] Hirose K, Murakami G, Minowa T, Kura H, Yamashita T. Lateral ligament injury of the ankle and associated articular cartilage degeneration in the talocrural joint: anatomic study using elderly cadavers. J Orthop Sci. 2004;9(1):37-43. doi: 10.1007/s00776-003-0732-9. PMID 14767703
- [Background] Kotlarz H, Gunnarsson CL, Fang H, Rizzo JA. Insurer and out-of-pocket costs of osteoarthritis in the US: evidence from national survey data. Arthritis Rheum. 2009 Dec;60(12):3546-53. doi: 10.1002/art.24984. PMID 19950287
- [Background] Verhagen RA, de Keizer G, van Dijk CN. Long-term follow-up of inversion trauma of the ankle. Arch Orthop Trauma Surg. 1995;114(2):92-6. doi: 10.1007/BF00422833. PMID 7734241
- [Background] Global Health Risks: Mortality and Burden of Disease Attributable to Selected Major RIsks. Geneva: World Health Organization; 2012
- [Background] Wester JU, Jespersen SM, Nielsen KD, Neumann L. Wobble board training after partial sprains of the lateral ligaments of the ankle: a prospective randomized study. J Orthop Sports Phys Ther. 1996 May;23(5):332-6. doi: 10.2519/jospt.1996.23.5.332. PMID 8728532
- [Background] Osborne MD, Rizzo TD Jr. Prevention and treatment of ankle sprain in athletes. Sports Med. 2003;33(15):1145-50. doi: 10.2165/00007256-200333150-00005. PMID 14719982
- [Background] Clark VM, Burden AM. A 4-week wobble board exercise programme imploved muscle onset latency and perceived stability in individuals with a functionally unstable ankle. Phys Ther Sport. 2005;6(4):181-187
- [Background] Dinesha A, Prasad B A. Effect of 2-week and 4-week wobble board exercise programme for improving the muscle onset latency and perceived stability in basketball players with recurrent ankle sprain. Indian J Physiother Occup Ther. 2011;5(1):27-32.
- [Background] Lee AJ, Lin WH. Twelve-week biomechanical ankle platform system training on postural stability and ankle proprioception in subjects with unilateral functional ankle instability. Clin Biomech (Bristol). 2008 Oct;23(8):1065-72. doi: 10.1016/j.clinbiomech.2008.04.013. Epub 2008 Jul 14. PMID 18621453
- [Background] Hoffman M, Payne VG. The effects of proprioceptive ankle disk training on healthy subjects. J Orthop Sports Phys Ther. 1995 Feb;21(2):90-3. doi: 10.2519/jospt.1995.21.2.90. PMID 7711762
- [Background] Soderberg GL, Cook TM, Rider SC, Stephenitch BL. Electromyographic activity of selected leg musculature in subjects with normal and chronically sprained ankles performing on a BAPS board. Phys Ther. 1991 Jul;71(7):514-22. doi: 10.1093/ptj/71.7.514. PMID 2052630
- [Background] Tropp H, Askling C, Gillquist J. Prevention of ankle sprains. Am J Sports Med. 1985 Jul-Aug;13(4):259-62. doi: 10.1177/036354658501300408. PMID 3927758
- [Background] Wright CJ, Linens SW, Cain MS. A Randomized Controlled Trial Comparing Rehabilitation Efficacy in Chronic Ankle Instability. J Sport Rehabil. 2017 Jul;26(4):238-249. doi: 10.1123/jsr.2015-0189. Epub 2016 Aug 24. PMID 27632874
- [Background] Cain MS, Garceau SW, Linens SW. Effects of a 4-Week Biomechanical Ankle Platform System Protocol on Balance in High School Athletes With Chronic Ankle Instability. J Sport Rehabil. 2017 Jan;26(1):1-7. doi: 10.1123/jsr.2015-0045. Epub 2016 Aug 24. PMID 27632846
- [Background] Stracciolini A, Casciano R, Levey Friedman H, Meehan WP 3rd, Micheli LJ. Pediatric sports injuries: an age comparison of children versus adolescents. Am J Sports Med. 2013 Aug;41(8):1922-9. doi: 10.1177/0363546513490644. Epub 2013 Jun 5. PMID 23739684
- [Background] Hogan KA, Gross RH. Overuse injuries in pediatric athletes. Orthop Clin North Am. 2003 Jul;34(3):405-15. doi: 10.1016/s0030-5898(03)00006-3. PMID 12974490
- [Background] Adirim TA, Cheng TL. Overview of injuries in the young athlete. Sports Med. 2003;33(1):75-81. doi: 10.2165/00007256-200333010-00006. PMID 12477379
- [Background] Kennedy JG, Hodgkins CW, Sculco P, Carter T, Robinson SP. Sports Injuries of The Foot and Ankle in The Adolescent Athlete. Int Sports Med J. 2006;7(2):85-97
- [Background] Stracciolini A, Casciano R, Friedman HL, Meehan WP 3rd, Micheli LJ. A closer look at overuse injuries in the pediatric athlete. Clin J Sport Med. 2015 Jan;25(1):30-5. doi: 10.1097/JSM.0000000000000105. PMID 24926911
- [Background] Malanga GA, Ramirez-Del Toro JA. Common injuries of the foot and ankle in the child and adolescent athlete. Phys Med Rehabil Clin N Am. 2008 May;19(2):347-71, ix. doi: 10.1016/j.pmr.2007.11.003. PMID 18395652
- [Background] Sobhani S, Dekker R, Postema K, Dijkstra PU. Epidemiology of ankle and foot overuse injuries in sports: A systematic review. Scand J Med Sci Sports. 2013 Dec;23(6):669-86. doi: 10.1111/j.1600-0838.2012.01509.x. Epub 2012 Jul 30. PMID 22846101
- [Background] Chambers HG. Ankle and foot disorders in skeletally immature athletes. Orthop Clin North Am. 2003 Jul;34(3):445-59. doi: 10.1016/s0030-5898(03)00031-2. PMID 12974494
- [Background] Damore DT, Metzl JD, Ramundo M, Pan S, Van Amerongen R. Patterns in childhood sports injury. Pediatr Emerg Care. 2003 Apr;19(2):65-7. doi: 10.1097/00006565-200304000-00001. PMID 12698027
- [Background] Swenson DM, Collins CL, Fields SK, Comstock RD. Epidemiology of U.S. high school sports-related ligamentous ankle injuries, 2005/06-2010/11. Clin J Sport Med. 2013 May;23(3):190-6. doi: 10.1097/JSM.0b013e31827d21fe. PMID 23328403
- [Background] Freeman MA. Instability of the foot after injuries to the lateral ligament of the ankle. J Bone Joint Surg Br. 1965 Nov;47(4):669-77. No abstract available. PMID 5846766
- [Background] Hertel J. Functional instability following lateral ankle sprain. Sports Med. 2000 May;29(5):361-71. doi: 10.2165/00007256-200029050-00005. PMID 10840868
- [Background] Tropp H. Commentary: Functional Ankle Instability Revisited. J Athl Train. 2002 Dec;37(4):512-515. No abstract available. PMID 12937576
- [Background] Bonnel F, Toullec E, Mabit C, Tourne Y; Sofcot. Chronic ankle instability: biomechanics and pathomechanics of ligaments injury and associated lesions. Orthop Traumatol Surg Res. 2010 Jun;96(4):424-32. doi: 10.1016/j.otsr.2010.04.003. Epub 2010 May 20. PMID 20493797
- [Background] Kavanagh JJ, Bisset LM, Tsao H. Deficits in reaction time due to increased motor time of peroneus longus in people with chronic ankle instability. J Biomech. 2012 Feb 2;45(3):605-8. doi: 10.1016/j.jbiomech.2011.11.056. Epub 2011 Dec 16. PMID 22177674
- [Background] McLeod MM, Gribble PA, Pietrosimone BG. Chronic Ankle Instability and Neural Excitability of the Lower Extremity. J Athl Train. 2015 Aug;50(8):847-53. doi: 10.4085/1062-6050-50.4.06. Epub 2015 Jun 19. PMID 26090710
- [Background] McVey ED, Palmieri RM, Docherty CL, Zinder SM, Ingersoll CD. Arthrogenic muscle inhibition in the leg muscles of subjects exhibiting functional ankle instability. Foot Ankle Int. 2005 Dec;26(12):1055-61. doi: 10.1177/107110070502601210. PMID 16390639
- [Background] McKeon PO, Hertel J. Spatiotemporal postural control deficits are present in those with chronic ankle instability. BMC Musculoskelet Disord. 2008 Jun 2;9:76. doi: 10.1186/1471-2474-9-76. PMID 18518994
- [Background] Feger MA, Donovan L, Hart JM, Hertel J. Lower extremity muscle activation in patients with or without chronic ankle instability during walking. J Athl Train. 2015 Apr;50(4):350-7. doi: 10.4085/1062-6050-50.2.06. Epub 2015 Jan 6. PMID 25562453
- [Background] Mitchell A, Dyson R, Hale T, Abraham C. Biomechanics of ankle instability. Part 1: Reaction time to simulated ankle sprain. Med Sci Sports Exerc. 2008 Aug;40(8):1515-21. doi: 10.1249/mss.0b013e31817356b6. PMID 18705024
- [Background] Mitchell A, Dyson R, Hale T, Abraham C. Biomechanics of ankle instability. Part 2: Postural sway-reaction time relationship. Med Sci Sports Exerc. 2008 Aug;40(8):1522-8. doi: 10.1249/MSS.0b013e31817356d6. PMID 18614937
- [Background] Brown CN, Mynark R. Balance deficits in recreational athletes with chronic ankle instability. J Athl Train. 2007 Jul-Sep;42(3):367-73. PMID 18059992
- [Background] Brown C, Bowser B, Simpson KJ. Movement variability during single leg jump landings in individuals with and without chronic ankle instability. Clin Biomech (Bristol). 2012 Jan;27(1):52-63. doi: 10.1016/j.clinbiomech.2011.07.012. Epub 2011 Aug 20. PMID 21862188
- [Background] Hubbard-Turner T, Turner MJ. Physical Activity Levels in College Students With Chronic Ankle Instability. J Athl Train. 2015 Jul;50(7):742-7. doi: 10.4085/1062-6050-50.3.05. Epub 2015 Apr 21. PMID 25898110
- [Background] Martin RL, Irrgang JJ, Burdett RG, Conti SF, Van Swearingen JM. Evidence of validity for the Foot and Ankle Ability Measure (FAAM). Foot Ankle Int. 2005 Nov;26(11):968-83. doi: 10.1177/107110070502601113. PMID 16309613
- [Background] Martin RL, Burdett RG. Development of the Foot and Ankle Disability Index (FADI) [Abstract]. J Orthop Sports Phys Ther. 1999;29:A32-A33
- [Background] Martin RL, Irrgang JJ. A survey of self-reported outcome instruments for the foot and ankle. J Orthop Sports Phys Ther. 2007 Feb;37(2):72-84. doi: 10.2519/jospt.2007.2403. PMID 17366962
- [Background] Hale SA, Hertel J. Reliability and Sensitivity of the Foot and Ankle Disability Index in Subjects With Chronic Ankle Instability. J Athl Train. 2005 Mar;40(1):35-40. PMID 15902322
- [Background] Carcia CR, Martin RL, Drouin JM. Validity of the Foot and Ankle Ability Measure in athletes with chronic ankle instability. J Athl Train. 2008 Apr-Jun;43(2):179-83. doi: 10.4085/1062-6050-43.2.179. PMID 18345343
- [Background] Docherty CL, Gansneder BM, Arnold BL, Hurwitz SR. Development and reliability of the ankle instability instrument. J Athl Train. 2006 Apr-Jun;41(2):154-8. PMID 16791299
- [Background] Hiller CE, Refshauge KM, Bundy AC, Herbert RD, Kilbreath SL. The Cumberland ankle instability tool: a report of validity and reliability testing. Arch Phys Med Rehabil. 2006 Sep;87(9):1235-41. doi: 10.1016/j.apmr.2006.05.022. PMID 16935061
- [Background] Wright CJ, Arnold BL, Ross SE, Linens SW. Recalibration and validation of the Cumberland Ankle Instability Tool cutoff score for individuals with chronic ankle instability. Arch Phys Med Rehabil. 2014 Oct;95(10):1853-9. doi: 10.1016/j.apmr.2014.04.017. Epub 2014 May 9. PMID 24814563
- [Background] Donahue M, Simon J, Docherty CL. Critical review of self-reported functional ankle instability measures. Foot Ankle Int. 2011 Dec;32(12):1140-6. doi: 10.3113/FAI.2011.1140. PMID 22381198
- [Background] Simon J, Donahue M, Docherty C. Development of the Identification of Functional Ankle Instability (IdFAI). Foot Ankle Int. 2012 Sep;33(9):755-63. doi: 10.3113/FAI.2012.0755. PMID 22995264
- [Background] Donahue M, Simon J, Docherty C. Reliability and Validity of a New Questionnaire Created to Establish the Presence of Functional Ankle Instability: The IdFAI. Athl Train Sports Health Care. 2013;5(1):38-43.
- [Background] Simon J, Donahue M, Docherty CL. Critical review of self-reported functional ankle instability measures: a follow up. Phys Ther Sport. 2014 May;15(2):97-100. doi: 10.1016/j.ptsp.2013.03.005. Epub 2013 Jul 25. PMID 23890746
- [Background] Riemann BL, Guskiewicz KM, Shields EW. Relationship Between Clinical and Forceplate Measures of Postural Stability. J Sport Rehabil. 1999;8(2):71-82.
- [Background] Docherty CL, Valovich McLeod TC, Shultz SJ. Postural control deficits in participants with functional ankle instability as measured by the balance error scoring system. Clin J Sport Med. 2006 May;16(3):203-8. doi: 10.1097/00042752-200605000-00003. PMID 16778539
- [Background] Linens SW, Ross SE, Arnold BL, Gayle R, Pidcoe P. Postural-stability tests that identify individuals with chronic ankle instability. J Athl Train. 2014 Jan-Feb;49(1):15-23. doi: 10.4085/1062-6050-48.6.09. Epub 2013 Dec 30. PMID 24377958
- [Background] Dobo B, White A, Linens S. Balance Error Scoring System Stances That Identify Division I Athletes With Chronic Ankle Instability Most in Need of Rehabilitation. Athl Train Sports Health Care. 2015;7(5):190-196
- [Background] McLeod TC, Armstrong T, Miller M, Sauers JL. Balance improvements in female high school basketball players after a 6-week neuromuscular-training program. J Sport Rehabil. 2009 Nov;18(4):465-81. doi: 10.1123/jsr.18.4.465. PMID 20108849
- [Background] Chrintz H, Falster O, Roed J. Single-leg Postural Equilibrium Test. Scand J Med Sci Sports. 1991;1(4):244-246
- [Background] Hiller CE, Refshauge KM, Herbert RD, Kilbreath SL. Balance and recovery from a perturbation are impaired in people with functional ankle instability. Clin J Sport Med. 2007 Jul;17(4):269-75. doi: 10.1097/JSM.0b013e3180f60b12. PMID 17620780
- [Background] Hertel J, Olmsted-Kramer LC. Deficits in time-to-boundary measures of postural control with chronic ankle instability. Gait Posture. 2007 Jan;25(1):33-9. doi: 10.1016/j.gaitpost.2005.12.009. Epub 2006 Jan 30. PMID 16446093
- [Background] Alsalaheen B, Haines J, Yorke A, Broglio SP. Reliability and Construct Validity of Limits of Stability Test in Adolescents Using a Portable Forceplate System. Arch Phys Med Rehabil. 2015 Dec;96(12):2194-200. doi: 10.1016/j.apmr.2015.08.418. Epub 2015 Aug 29. PMID 26325240
- [Background] Docherty CL, Arnold BL, Gansneder BM, Hurwitz S, Gieck J. Functional-Performance Deficits in Volunteers With Functional Ankle Instability. J Athl Train. 2005 Mar;40(1):30-34. PMID 15902321
- [Background] Chambers RB, Cook TM, Cowell HR. Surgical reconstruction for calcaneonavicular coalition. Evaluation of function and gait. J Bone Joint Surg Am. 1982 Jul;64(6):829-36. PMID 6806302
- [Background] Buchanan AS, Docherty CL, Schrader J. Functional performance testing in participants with functional ankle instability and in a healthy control group. J Athl Train. 2008 Jul-Aug;43(4):342-6. doi: 10.4085/1062-6050-43.4.342. PMID 18668180
- [Background] Eechaute C, Vaes P, Duquet W. Functional performance deficits in patients with CAI: validity of the multiple hop test. Clin J Sport Med. 2008 Mar;18(2):124-9. doi: 10.1097/JSM.0b013e31816148d2. PMID 18332686
- [Background] Eechaute C, Vaes P, Duquet W. The dynamic postural control is impaired in patients with chronic ankle instability: reliability and validity of the multiple hop test. Clin J Sport Med. 2009 Mar;19(2):107-14. doi: 10.1097/JSM.0b013e3181948ae8. PMID 19451764
- [Background] Munn J, Beard DJ, Refshauge KM, Lee RW. Do Functional-Performance Tests Detect Impairment in Subjects With Ankle Instability. J Sport Rehabil. 2002;11(1):40-50.
- [Background] Noyes FR, Barber SD, Mangine RE. Abnormal lower limb symmetry determined by function hop tests after anterior cruciate ligament rupture. Am J Sports Med. 1991 Sep-Oct;19(5):513-8. doi: 10.1177/036354659101900518. PMID 1962720
- [Background] Barber SD, Noyes FR, Mangine RE, McCloskey JW, Hartman W. Quantitative assessment of functional limitations in normal and anterior cruciate ligament-deficient knees. Clin Orthop Relat Res. 1990 Jun;(255):204-14. PMID 2347154
- [Background] Olmsted LC, Carcia CR, Hertel J, Shultz SJ. Efficacy of the Star Excursion Balance Tests in Detecting Reach Deficits in Subjects With Chronic Ankle Instability. J Athl Train. 2002 Dec;37(4):501-506. PMID 12937574
- [Background] Hertel J, Braham RA, Hale SA, Olmsted-Kramer LC. Simplifying the star excursion balance test: analyses of subjects with and without chronic ankle instability. J Orthop Sports Phys Ther. 2006 Mar;36(3):131-7. doi: 10.2519/jospt.2006.36.3.131. PMID 16596889
- [Background] Gribble PA, Hertel J. Considerations for normalizing measures of the star excursion balance test. Meas Phys Educ Exerc Sci. 2003;7(2):89-100.
- [Background] Robinson RH, Gribble PA. Support for a reduction in the number of trials needed for the star excursion balance test. Arch Phys Med Rehabil. 2008 Feb;89(2):364-70. doi: 10.1016/j.apmr.2007.08.139. PMID 18226664
- [Background] Hertel J, Miller SJ, Denegar CR. Intratester and intertester reliability during the star excursion balance tests. J Sports Rehabil. 2000;9(2):104-116.
- [Background] Hubbard TJ, Kramer LC, Denegar CR, Hertel J. Contributing factors to chronic ankle instability. Foot Ankle Int. 2007 Mar;28(3):343-54. doi: 10.3113/FAI.2007.0343. PMID 17371658
- [Background] Plisky PJ, Gorman PP, Butler RJ, Kiesel KB, Underwood FB, Elkins B. The reliability of an instrumented device for measuring components of the star excursion balance test. N Am J Sports Phys Ther. 2009 May;4(2):92-9. PMID 21509114
- [Background] Plisky PJ, Rauh MJ, Kaminski TW, Underwood FB. Star Excursion Balance Test as a predictor of lower extremity injury in high school basketball players. J Orthop Sports Phys Ther. 2006 Dec;36(12):911-9. doi: 10.2519/jospt.2006.2244. PMID 17193868
- [Background] Hertel J. Sensorimotor deficits with ankle sprains and chronic ankle instability. Clin Sports Med. 2008 Jul;27(3):353-70, vii. doi: 10.1016/j.csm.2008.03.006. PMID 18503872
- [Background] Gribble PA, Hertel J, Plisky P. Using the Star Excursion Balance Test to assess dynamic postural-control deficits and outcomes in lower extremity injury: a literature and systematic review. J Athl Train. 2012 May-Jun;47(3):339-57. doi: 10.4085/1062-6050-47.3.08. PMID 22892416
- [Background] Mattacola CG, Dwyer MK. Rehabilitation of the Ankle After Acute Sprain or Chronic Instability. J Athl Train. 2002 Dec;37(4):413-429. PMID 12937563
- [Background] Eils E, Rosenbaum D. A multi-station proprioceptive exercise program in patients with ankle instability. Med Sci Sports Exerc. 2001 Dec;33(12):1991-8. doi: 10.1097/00005768-200112000-00003. PMID 11740289
- [Background] Hale SA, Hertel J, Olmsted-Kramer LC. The effect of a 4-week comprehensive rehabilitation program on postural control and lower extremity function in individuals with chronic ankle instability. J Orthop Sports Phys Ther. 2007 Jun;37(6):303-11. doi: 10.2519/jospt.2007.2322. PMID 17612356
- [Background] Lee KY, Lee HJ, Kim SE, Choi PB, Song SH, Jee YS. Short term rehabilitation and ankle instability. Int J Sports Med. 2012 Jun;33(6):485-96. doi: 10.1055/s-0032-1301933. Epub 2012 Mar 15. PMID 22422307
- [Background] Soligard T, Myklebust G, Steffen K, Holme I, Silvers H, Bizzini M, Junge A, Dvorak J, Bahr R, Andersen TE. Comprehensive warm-up programme to prevent injuries in young female footballers: cluster randomised controlled trial. BMJ. 2008 Dec 9;337:a2469. doi: 10.1136/bmj.a2469. PMID 19066253
- [Background] Emery CA, Rose MS, McAllister JR, Meeuwisse WH. A prevention strategy to reduce the incidence of injury in high school basketball: a cluster randomized controlled trial. Clin J Sport Med. 2007 Jan;17(1):17-24. doi: 10.1097/JSM.0b013e31802e9c05. PMID 17304001
- [Background] Emery CA, Meeuwisse WH. The effectiveness of a neuromuscular prevention strategy to reduce injuries in youth soccer: a cluster-randomised controlled trial. Br J Sports Med. 2010 Jun;44(8):555-62. doi: 10.1136/bjsm.2010.074377. PMID 20547668
- [Background] Docherty CL, Moore JH, Arnold BL. Effects of strength training on strength development and joint position sense in functionally unstable ankles. J Athl Train. 1998 Oct;33(4):310-4. PMID 16558526
- [Background] Kaminski TW, Buckley BD, Powers ME, Hubbard TJ, Ortiz C. Effect of strength and proprioception training on eversion to inversion strength ratios in subjects with unilateral functional ankle instability. Br J Sports Med. 2003;37(5):410-5; discussion 415. doi: 10.1136/bjsm.37.5.410. PMID 14514531
- [Background] Han K, Ricard MD, Fellingham GW. Effects of a 4-week exercise program on balance using elastic tubing as a perturbation force for individuals with a history of ankle sprains. J Orthop Sports Phys Ther. 2009 Apr;39(4):246-55. doi: 10.2519/jospt.2009.2958. PMID 19346625
- [Background] Hall EA, Docherty CL, Simon J, Kingma JJ, Klossner JC. Strength-training protocols to improve deficits in participants with chronic ankle instability: a randomized controlled trial. J Athl Train. 2015 Jan;50(1):36-44. doi: 10.4085/1062-6050-49.3.71. Epub 2014 Nov 3. PMID 25365134
- [Background] Osborne MD, Chou LS, Laskowski ER, Smith J, Kaufman KR. The effect of ankle disk training on muscle reaction time in subjects with a history of ankle sprain. Am J Sports Med. 2001 Sep-Oct;29(5):627-32. doi: 10.1177/03635465010290051601. PMID 11573922
- [Background] Linens SW, Ross SE, Arnold BL. Wobble Board Rehabilitation for Improving Balance in Ankles With Chronic Instability. Clin J Sport Med. 2016 Jan;26(1):76-82. doi: 10.1097/JSM.0000000000000191. PMID 25831410
- [Background] Emery CA, Cassidy JD, Klassen TP, Rosychuk RJ, Rowe BH. Effectiveness of a home-based balance-training program in reducing sports-related injuries among healthy adolescents: a cluster randomized controlled trial. CMAJ. 2005 Mar 15;172(6):749-54. doi: 10.1503/cmaj.1040805. PMID 15767608
- [Background] Wortmann MA, Docherty CL. Effect of balance training on postural stability in subjects with chronic ankle instability. J Sport Rehabil. 2013 May;22(2):143-9. doi: 10.1123/jsr.22.2.143. Epub 2012 Oct 30. PMID 23117258
- [Background] Gerber JP, Williams GN, Scoville CR, Arciero RA, Taylor DC. Persistent disability associated with ankle sprains: a prospective examination of an athletic population. Foot Ankle Int. 1998 Oct;19(10):653-60. doi: 10.1177/107110079801901002. PMID 9801078
- [Background] Marx RG, Stump TJ, Jones EC, Wickiewicz TL, Warren RF. Development and evaluation of an activity rating scale for disorders of the knee. Am J Sports Med. 2001 Mar-Apr;29(2):213-8. doi: 10.1177/03635465010290021601. PMID 11292048
- [Derived] Cain MS, Ban RJ, Chen YP, Geil MD, Goerger BM, Linens SW. Four-Week Ankle-Rehabilitation Programs in Adolescent Athletes With Chronic Ankle Instability. J Athl Train. 2020 Aug 1;55(8):801-810. doi: 10.4085/1062-6050-41-19. PMID 32577737